CLINICAL TRIAL: NCT03037281
Title: Does the Release Profile of Nociceptin From Immunocytes Differ in Healthy Volunteers and Critically Ill Patients With Sepsis?
Brief Title: Release of Nociceptin From Granulocytes in Sepsis
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: The Royal College of Anaesthetists (Other); University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0554
Record Dates: First submitted 2017-01-25; First posted 2017-01-31 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2019-04

CONDITIONS: Sepsis; Septic Shock; Sepsis Syndrome; Severe Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic: Patients admitted to the intensive care unit with a diagnosis of sepsis. For the purposes of this study, patients must have a diagnosis of sepsis; SIRS (2 of pulse >90, WCC, BP, Oxygen(Dellinger et al., 2013)) with microbiological evidence of infection (positive blood culture, urine dipstick, compatible history or examination, radiographic evidence)
  Interventions: Diagnostic Test: Septic
- Healthy volunteers: Healthy volunteers will be approached within the Department of Cardiovascular Sciences, and provided with the PIS, with consent taken by one of the investigating team.
  Interventions: Diagnostic Test: Septic

INTERVENTIONS:
Diagnostic Test: Septic — 30mls of blood will be sampled by venepuncture, or sampled from indwelling lines (in the case of septic patients on intensive care). Blood will be sampled using standard techniques, and transferred to EDTA containing blood bottles, and undergo processing immediately.
  Other Names: Healthy volunteers

SUMMARY:
Nociceptin is a protein found in the body, with a number of functions in the central nervous system, blood vessels and the gut. There is evidence that it may have a role in controlling the immune response to infection, and may act as a link between the brain and immune system.

In infection, or after surgery, there is an increase in nociceptin, and subjects greater elevations of nociceptin have a poorer outcome. There is evidence that cells of the immune system may produce nociceptin, although it is not yet known which cells are capable of producing it, and what "switches on" production.

This study aims to determine

1. Which cells of the immune system can produce nociceptin
2. If there is a difference in the ability to produce nociceptin between healthy volunteers and patients with severe infections

ELIGIBILITY:
Inclusion Criteria:

* For septic patients;

  1. Participant is willing and able to give informed consent for participation in the study, or if lacking capacity, a next of kin or advocate is willing and able to give assent for participation in the study. Must be able to read and understand English.
  2. Male or Female, aged 18 years or above.
  3. Diagnosed with sepsis and admitted to the intensive care unit.
  4. Able (in the Investigators opinion) and willing to comply with all study requirements.
  5. Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Healthy Volunteers;

1. Participant is willing and able to give informed consent for participation in the study. Must be able to read and understand English.
2. Male or Female, aged 18 years or above and be
3. In good health.
4. Have had no course of medication, whether prescribed or over-the-counter, in the four weeks before first study dose and no individual doses in the final two weeks other than mild analgesia, vitamins and mineral supplements or, for females, oral contraceptives
5. Able (in the Investigators opinion) and willing to comply with all study requirements.
6. Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* 1. Conditions which may make phlebotomy hazardous to the participant (such as significant bleeding disorders or anaemia, or allergy), or to the investigator (blood viral infection).

  2. Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

  3. Participants who have participated in another research study involving an investigational product in the past 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers - Adults, staff or students at the Univesity of Leicester, with no significant comorbidity Septic patients - Adult patients admitted to the adult intensive care unit, Leicester Royal Infirmary, with a diagnosis of sepsis
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Hebbes, BSc, Principal Investigator — University of Leicester
Locations (2):
- United Kingdom (2):
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - University of Leicester, Leicester, Leicestershire

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Septic | Healthy Volunteers
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Septic | Healthy Volunteers | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 5 | 8 | 13
Age, Continuous [Mean (Full Range); unit: years] | 75.5 [55 to 85] | 34.5 [26 to 47] | 52 [26 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responsive Biosensor Cells Responding to Granulocyte Addition in the Presence and Absence of NOP Antagonist
Description: Measure of N/OFQ presence in granulocytes and associated supernatant
Time Frame: Day 1
Population: Biosensor cells
Measure: Mean (Standard Deviation); unit: mean % responsive biosensor cells
Units Other Than Participants: Biosensor cells
Groups:
- Septic (+NOP Antagonist SB612111): Cells harvested from patients with sepsis, treated in an environment containing the NOP antagonist SB612111
- Septic (N/OFQ Control): Control treatment of biosensor cells with N/OFQ as a control
- Healthy Volunteers (+NOP Antagonist SB612111): Cells harvested from healthy volunteers in an environment containing the NOP antagonist SB612111
- Healthy Volunteers (N/OFQ Control): Cells taken from healthy volunteers treated with N/OFQ as a control
Arm/Group | Septic | Septic (+NOP Antagonist SB612111) | Septic (N/OFQ Control) | Healthy Volunteers | Healthy Volunteers (+NOP Antagonist SB612111) | Healthy Volunteers (N/OFQ Control)
Number analyzed (Participants) | 6 | 6 | 6 | 8 | 8 | 8
Number analyzed (Biosensor cells) | 138 | 40 | 258 | 210 | 184 | 410
mean % responsive biosensor cells
  Eosinophils | 34.25907426 (26.36477836) | 5.882352941 (NA) — Insufficient number of responsive cells as a fraction of overall number of cells extracted to allow SD to be calculated. | 44.17193917 (30.09734468) | 25.13095238 (31.52494693) | 17.86976912 (14.33561565) | 39.97303622 (32.13672569)
  Neutrophils | 25.73232323 (25.95276607) | 8.712121212 (0.535686955) | 48.66792929 (37.86453531) | 32.34442641 (22.5667298) | 12.87518038 (20.00326171) | 17.06777597 (15.88672067)

2. Secondary Outcome: Granulocyte Count
Description: Count of the number of neutrophils in the original sample
Time Frame: Day 1
Measure: Mean (Full Range); unit: x10^7 cells ml-1
Arm/Group | Septic | Healthy Volunteers
Number analyzed (Participants) | 6 | 8
x10^7 cells ml-1
  Neutrophils | 5.07 [3.33 to 6.4] | 2.05 [0.94 to 3.4]
  Eosinophils | 0.98 [0.4 to 1.9] | 1.61 [0.53 to 2.44]

3. Secondary Outcome: Mortality In-hospital, at 30 Days
Description: All cause mortality at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Septic | Healthy Volunteers
Number analyzed (Participants) | 6 | 8
Participants | 3 | 0

4. Secondary Outcome: Time to ICU Discharge (or Death if on ICU)
Time Frame: Time to ICU discharge (or death if on ICU)
Measure: Median (Full Range); unit: days
Arm/Group | Septic
Number analyzed (Participants) | 4
days | 7.5 [3 to 24]

5. Secondary Outcome: Time to Death or Discharge
Description: Time to death or discharge (days)
Time Frame: Number of days between admission and death or discharge from hospital
Measure: Median (Full Range); unit: days
Arm/Group | Septic
Number analyzed (Participants) | 6
days | 17.5 [3 to 59]

6. Secondary Outcome: Acute Physiology and Chronic Health Evaluation (APACHE-2) Score
Description: The Acute Physiology and Chronic Health Evaluation (APACHE-2) score for the patient.
  APACHE 2 is an international standard,12 variable score from 0-71 reflecting disease severity in the critically unwell during the first 24 hours of illness. The score is a combined measure of illness severity (acute physiology), and background chronic health factors. Increased score represents increased predicted mortality.
  Variables recorded include AaDO2 or PaO2 (depending on FiO2), temperature, mean arterial pressure, blood pH, heart rate, respiratory rate, serum sodium, serum potassium, creatinine, hematocrit, white blood cell count, Glasgow Coma Scale
  Knaus WA, Draper EA, Wagner DP, Zimmerman JE (1985). "APACHE II: a severity of disease classification system". Critical Care Medicine. 13 (10): 818-29
Time Frame: Day 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Septic
Number analyzed (Participants) | 6
score on a scale | 19.8 [6 to 31]

7. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Score
Description: The Sequential Organ Failure Assessment (SOFA) score for the patient, a score predictive of mortality in sepsis for intensive care patients based on respiratory, cardiovascular, hepatic, coagulation, renal and neurological function (each scored 0-4, with a maximum overall score of 24). The worst (most deranged) physiological values for the first 24 hours are used. A higher score predicts increased mortality. The mortality breakdown for each sofa score range is - SOFA 0-6 (<10% mortality), 7-9 (15-20%), 10-12 (40-50%), 13-14 (50 - 60%), 15 (> 80%), 16 to 24 (> 90%)
Time Frame: Day 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Septic
Number analyzed (Participants) | 6
score on a scale | 9.33 [5 to 12]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Septic | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 3/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

LIMITATIONS AND CAVEATS:
Technical problems with both measurement and immunocyte extraction contributed to high variability with the assay and inconsistencies.Small numbers of subjects recruited precluded robust statistical analysis.Basophil extraction very low - not viable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT03037281/Prot_SAP_000.pdf